CLINICAL TRIAL: NCT04856644
Title: Evaluation of the Efficacy and Safety of a Short-course, Daily, 4-month Regimen Including Isoniazid, Pyrazinamide, Rifapentine and Moxifloxacin (2HZPM/2HPM) for the Treatment of Drug-susceptible Pulmonary Tuberculosis in Taiwan (ESCAPE-TB)
Brief Title: Evaluation of the Efficacy and Safety of a 4-month Daily Regimen (2HZPM/2HPM) for Treatment of Pulmonary TB
Acronym: ESCAPE-TB
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Collaborators: National Taiwan University (Other); Taipei Veterans General Hospital, Taiwan (Other Government); Chang Gung Memorial Hospital (Other); Centers for Disease Control, Taiwan (Other Government)
Responsible Party: Principal Investigator, Susan Shin-Jung Lee, Attending physiciian, Division of Infectious Diseases, Kaohsiung Veterans General Hospital.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KSVGH21-CT5-49
Record Dates: First submitted 2021-03-31; First posted 2021-04-23 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Tuberculosis, Pulmonary
MeSH Terms: conditions — Tuberculosis, Pulmonary | interventions — rifapentine; Moxifloxacin

STUDY DESIGN:
Intervention Model Description: The intervention group: all patients recruited into the study will receive the 4-month regimen The comparator group: historical control in those who received the standard 6-month regimen
Masking Description: Masking will not be done
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 4-month regimen (2HZPM/2HPM) (Experimental): * Eight weeks of daily treatment with isoniazid (H), pyrazinamide (Z), rifapentine (P), and moxifloxacin (M), followed by
  * Nine weeks of daily treatment with isoniazid, rifapentine and moxifloxacin
  Interventions: Drug: 4-month rifapentine-based regimen
- Standard 6-month regimen (2HERZ/4HR) historical control (No Intervention): a standard, six-month regimen, with
  * Eight weeks of daily treatment with isoniazid (H), rifampin (R), pyrazinamide (Z) and ethambutol (E) followed by
  * Eighteen weeks of daily treatment with isoniazid and rifampin, with or without ethambutol

INTERVENTIONS:
Drug: 4-month rifapentine-based regimen — 8 weeks of isoniazid, pyrazinamide, rifapentine, and moxifloxacin, followed by 9 weeks of isoniazid, rifapentine and moxifloxacin
  Other Names: rifapentine; moxifloxacin; priftin
  Arms: 4-month regimen (2HZPM/2HPM)

SUMMARY:
The development of efficacious, safe, and shorter treatment regimens could significantly improve TB management and treatment success rates. This prospective, 3-year, single arm study is to evaluate the efficacy and safety of a short-course, 4-month regimen including isoniazid(H), pyrazinamide(P), rifapentine (P), and moxifloxacin(M) (2HZPM/2HPM) for the treatment of drug-susceptible, pulmonary tuberculosis, and compared with a historical control group receiving the standard six-month regimen.

DETAILED DESCRIPTION:
Shorter regimens have the potential to impact on TB control by reducing TB incidence and mortality, and improve outcomes by increasing patient adherence to treatments and decreasing duration to cure, in addition to reducing costs to the health system and the patient. The purpose of this prospective, three year, single arm study is to evaluate whether a short course, four-month regimen containing rifapentine and moxifloxacin (2HZPM/2HPM) are as effective and/or as tolerable as the standard six-month regimen for the treatment of drug-susceptible, pulmonary tuberculosis (TB). A historical group receiving the standard six-month regimen is used as control at a ratio of 1:2. The pharmacokinetic and pharmacodynamic profile of rifapentine in Asian patients. Analysis of of histocompatibility leucocyte antigen (HLA) associations with adverse events and changes in biomarkers will be done.

ELIGIBILITY:
Inclusion Criteria:

1. Suspected newly diagnosed pulmonary TB plus one of the following: a) at least one sputum specimen positive for acid-fast bacilli on smear microscopy OR b) at least one sputum specimen positive for Mycobacterium tuberculosis by culture or "Gene Xpert MTB/RIF" testing, with rifamycin resistance not detected, OR c) histopathologic findings compatible with mycobacterial infection including a positive acid-fast stain
2. Patient with a history of being untreated for 3 years after cure from a previous episode of TB can be included.
3. Age 20 years or older
4. For women of childbearing potential, a negative pregnancy test at or within seven (7) days prior to screening is required, and must agree to practice a barrier method of contraception during study drug treatment, or be surgically sterilized or have an intrauterine contraceptive device in place.
5. Laboratory parameters performed at or within 14 days prior to enrollment:

   * Serum or plasma alanine aminotransferase (ALT) less than or equal to 3 times the upper limit of normal
   * Serum or plasma total bilirubin less than or equal to 2.5 times the upper limit of normal
   * Serum or plasma creatinine level less than or equal to 2 times the upper limit of normal or Creatinine clearance (CrCl) level greater than 30 mL/min.
   * Serum or plasma potassium level greater than or equal to 3.5 milliequivalent/L
   * Hemoglobin level of 7.0 g/dL or greater
   * Platelet count of 100,000/mm3 or greater
6. Patient signed a written informed consent

Exclusion Criteria:

1. Pregnant or breast-feeding.
2. Unable to take oral medications.
3. Previously enrolled in this study.
4. Received any investigational drug in the past 3 months.
5. More than 14 days of systemic treatment with any antituberculous drugs preceding initiation of study drugs.
6. Known history of prolonged QT syndrome.
7. Suspected or documented TB involving the central nervous system and/or bones and/or joints, and/or miliary tuberculosis and/or pericardial tuberculosis.
8. Weight less than 40.0 kg.
9. Known allergy or intolerance to any of the study medications.
10. Individuals will be excluded from enrollment if, at the time of enrollment, their M. tuberculosis isolate is already known to be resistant to any one or more of the following: rifampin, isoniazid, pyrazinamide, ethambutol, or fluoroquinolones.
11. Medical conditions, including HIV infection and others conditions that, in the investigator's judgment, make study participation not in the individual's best interest.
12. Late exclusions: Drug-resistant TB by either rapid sputum based test (Gene Expert) or resistance testing using an indirect susceptibility test in liquid culture to isoniazid, rifampin, ethambutol, pyrazinamide or resistance to moxifloxacin or rifapentine by microdilution agar proportion test.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 333 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
TB disease free survival at 12 months | 12 months after study treatment assignment
  Number and follow up time of participants without TB disease at 12 months after study treatment assignment in person-months
Grade 3 or higher adverse events during study drug treatment | 0-4 months
  The number of participants with grade 3 or higher adverse events during study drug treatment divided by total number of participants

SECONDARY OUTCOMES:
Early sterilizing activity (Negative sputum cultures at end of intensive 8 weeks phase) | 8 weeks
  The number of patients with a negative sputum culture at the end of intensive phase therapy at 8 weeks divided by total number of participants
Time to stable sputum conversion (Time in days from conversion of a positive sputum culture to negative sputum culture) | 4, 8, 12, 17 weeks, 6 months, 12 months
  Number of days from start of treatment to first negative sputum culture that remain negative thereafter
Speed of decline of sputum viable bacilli by automated mycobacteria growth indicator tube (MGIT) days to detection | 2-8 weeks
  Number of days from loading of sputum culture into MGIT to the day of detection of viable mycobacteria
TB disease-free survival at 12 months after study treatment assignment assuming all losses to follow-up and non-TB deaths have an unfavorable outcome (Sensitivity analyses assuming all losses to follow-up and non-TB deaths have an unfavorable outcome) | 12 months
  Number and follow up time of participants without TB disease at 12 months after study treatment assignment assuming all losses to follow-up and non-TB deaths have an unfavorable outcome (Sensitivity analyses assuming all losses to follow-up and non-TB deaths have an unfavorable outcome) in person-months
TB disease-free survival at 12 months after study treatment assignment assuming all losses to follow-up and non-TB deaths have an favorable outcome (Sensitivity analyses assuming all losses to follow-up and non-TB deaths have an favorable outcome) | 12 months
  Number and follow up time of participants without TB disease at 12 months after study treatment assignment assuming all losses to follow-up and non-TB deaths have an favorable outcome (Sensitivity analyses assuming all losses to follow-up and non-TB deaths have an favorable outcome) in person-months
Rates of treatment discontinuation for reasons other than ineligibility (late exclusions due to drug resistance or HIV status) | 0-4 months
  Number of participants who discontinued treatment for reasons other than ineligibility (late exclusions due to drug resistance or HIV status) divided by total number of participants
All-cause mortality at 4 months post-treatment assignment | 4 months
  Number of participants who died at 4 months divided by number of participants
All-cause mortality at 12 months post-treatment assignment | 12 months
  Number of participants who died at 12 months divided by number of participants
Attributable mortality at 4 months post-treatment assignment | 4 months
  Number of patients who died due to reasons attributable to tuberculosis at 4 months post-treatment assignment divided by number of participants
Attributable mortality at 12 months post-treatment assignment | 12 months
  Number of patients who died due to reasons attributable to tuberculosis at 12 months post-treatment assignment divided by number of participants
Changes in interferon-gamma levels during treatment compared to baseline | 2, 4, 8, 12 weeks
  interferon-gamma levels during treatment minus baseline levels
Changes in tumor necrosis factor-alpha levels during treatment compared to baseline | 2, 4, 8, 12 weeks
  Tumor necrosis factor-alpha levels during treatment minus baseline levels
Changes in interleukin-12 and interleukin-6 levels during treatment compared to baseline | 2, 4, 8, 12 weeks
  Interleukin-12 levels during treatment minus baseline levels
Changes in triggering receptor expressed on myeloid cells-1 (TREM-1) levels during treatment compared to baseline | 2, 4, 8, 12 weeks
  Triggering receptor expressed on myeloid cells-1 (TREM-1) levels during treatment minus baseline levels

OTHER OUTCOMES:
HLA Genotyping to detect predictors for occurrence of severe drug adverse events including skin rash and hepatitis. | 0-4 months
  Identify HLA genotypes associated with severe drug adverse events such as greater than grade 2 hepatitis and/or skin rash
Maximum plasma concentration (Cmax) of rifapentine | 0, 2, 4, 8, 12 weeks
  Serum concentration of rifapentine by determining area under the curve

CONTACTS AND LOCATIONS:
Overall Officials: Susan Shin-Jung Lee, M.D., Ph.D., Principal Investigator — Kaohsiung Veterans General Hospital.
Locations (4):
- Taiwan (4):
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Taipei Veterans General Hospital, Taipei
  - National Taiwan University Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan

IPD SHARING:
Plan to Share IPD: Undecided